CLINICAL TRIAL: NCT00766389
Title: Retinal Nerve Fiber Layer Thickness Analysis With Cirrus HD OCT Versus Stratus OCT
Brief Title: Retinal Nerve Fiber Layer Thickness Analysis With Cirrus HD OCT Versus Stratus Optical Coherence Tomography (OCT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Gong Je Seong, Yonsei University College of Medicine
Other Study IDs: 3-2008-0113
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Retinal nerve fiber layer; Cirrus OCT; Stratus OCT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Defined glaucoma patients
- 2: Glaucoma suspects and normal controls

SUMMARY:
The Cirrus HD OCT, a new spectral domain optical coherence tomography (OCT), has better resolution than the previous time domain Stratus OCT. Discriminating ability of these two OCTs for diagnosis of glaucoma and judgement of disease progression will be studied.

DETAILED DESCRIPTION:
The Cirrus HD OCT is a new spectral domain OCT. Even though its resolution and speed are much better than the previous time domain Stratus OCT, its diagnostic power for glaucoma detection and judgement of disease progression should be directly compared with Stratus OCT. In the present study, we will review the data of peripapillary retinal nerve fiber layer thickness measurement using the Cirrus HD OCT and Stratus OCT. Their discriminating ability for diagnosis of glaucoma and judgement of disease progression will be compared using the ROC curves and Cohen's kappa.

ELIGIBILITY:
Inclusion Criteria:

* Retinal nerve fiber layer analysis with Cirrus OCT and Stratus OCT within 1 month

Exclusion Criteria:

* Intraocular surgeries history
* DM
* High refractive error ( < -4.00 diopters, or > + 4.00 diopters)
* Media opacity

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Defined glaucoma patients and glaucoma suspects
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | When the OCT images are taking

SECONDARY OUTCOMES:
Visual field | When the OCT images are taking
Red-free fundus photo | When the OCT images are taking
Intraocular pressure | When the OCT images are taking
Central corneal thickness | When the OCT images are taking

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Study Chair — Yonsei University
Locations (1):
- Gong Je Seong, Seoul, South Korea